CLINICAL TRIAL: NCT03164317
Title: A Cluster Randomised Controlled Trial of M-health Enabled, Nurse Care Coordinator Led Intervention to Improve Management of Hypertension in India: m-Power Heart Project
Brief Title: To Test the Effectiveness of a Trained Nurse Led, M-health Enabled Intervention to Control Blood Pressure in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Chronic Disease Control, India (Other)
Collaborators: All India Institute of Medical Sciences (Other); Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr. Dorairaj Prabhakaran, Executive Director, Centre for Chronic Disease Control, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCDC-2017-001
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hypertension
Keywords: Hypertension; High blood pressure; Task shifting; Decision support system
MeSH Terms: conditions — Hypertension | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Trained NCC together with electronic decision support system
  Interventions: Other: Intervention
- Control (Other): No trained NCC and electronic decision support system
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — A trained nurse care coordinator enabled with a electronic decision support system placed at the CHCs to share the task of management of hypertension.
  Arms: Intervention
Other: Control — No NCC or EDSS will be placed in the CHCs. Doctors working in the CHCs will be given training (one day) on evidence based management of hypertension
  Arms: Control

SUMMARY:
This study evaluates the effect of a mobile health technology enabled trained nurse led intervention on control of blood pressure among patients with hypertension seeking care in the community health centres in the southern state of Andhra Pradesh, India. half the community health centres will receive the intervention and the other half will receive the routine care.

DETAILED DESCRIPTION:
The burden of hypertension is very high in India but the control rates of hypertension are very low. One of the important reasons for this is the lack of awareness and the inability of the doctors working in busy out patient settings of public health facilities to care adequately for the patients. Hence there is a need for task shifting.

In this trial a trained nurse care coordinator will be placed in the Community Health Centres (CHCs) and she will be provided with an Electronic Decision Support System (EDSS), in the form of an android application installed on a tablet, to treat hypertension. The trial will be carried out in twelve CHCs of Visakhapatnam district in southern Indian state of Andhra Pradesh.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged ≥30 years.
2. Willing to provide written informed consent for the study.
3. Identified as suffering from hypertension (≥160/100 mmHg) with or without co-morbidities such as left ventricular hypertrophy, heart failure, coronary artery disease, peripheral vascular disease, or diabetes mellitus

Exclusion Criteria:

1. Participants aged <30years
2. Unwilling/unable to provide written informed consent for the study
3. Having malignancies or life threatening conditions
4. Currently participating in other clinical trials
5. Those with plans to move residence in the year ahead.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1872 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Difference in the mean systolic blood pressure | 12 months
  Difference in the mean systolic blood pressure between the intervention and control arm at the end of the intervention

SECONDARY OUTCOMES:
Compliance to therapy | 12 months
  Difference in compliance to therapy from baseline to one year between the intervention and control arm
Follow up with the physician | 12 months
  Difference in follow up rate from baseline to one year between the intervention and control arm

CONTACTS AND LOCATIONS:
Overall Officials: Dorairaj Prabhakaran, MD, DM, Principal Investigator — Centre for Chronic Disease Control
Locations (12):
- India (12):
  - Community Health Centre, Aganampudi, Andhra Pradesh
  - Area Hospital, Anakapalle, Andhra Pradesh
  - Community Health Centre, Araku, Andhra Pradesh
  - Community Health Centre, Bhimili, Andhra Pradesh
  - Community Health Centre, Chintapalli, Andhra Pradesh
  - Community Health Centre, Chodavaram, Andhra Pradesh
  - Community Health Centre, K Kotpadu, Andhra Pradesh
  - Community Health Centre, Kotavaratla, Andhra Pradesh
  - Community Health Centre, Nakkapalli, Andhra Pradesh
  - Community Health Centre, Pāderu, Andhra Pradesh
  - Community Health Centre, V Madugula, Andhra Pradesh
  - Community Health Centre, Yelamanchili, Andhra Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srinivasapura Venkateshmurthy N, Mc Namara K, Koorts H, Mohan S, S Ajay V, Jindal D, Malipeddi BR, Roy A, Tandon N, Prabhakaran D, Worsley T, Maddison R, O'Reilly S. Process evaluation protocol for a cluster randomised trial of a complex, nurse-led intervention to improve hypertension management in India. BMJ Open. 2019 May 19;9(5):e027841. doi: 10.1136/bmjopen-2018-027841. PMID 31110103
- [Derived] Srinivasapura Venkateshmurthy N, Ajay VS, Mohan S, Jindal D, Anand S, Kondal D, Tandon N, Rao MB, Prabhakaran D. m-Power Heart Project - a nurse care coordinator led, mHealth enabled intervention to improve the management of hypertension in India: study protocol for a cluster randomized trial. Trials. 2018 Aug 7;19(1):429. doi: 10.1186/s13063-018-2813-2. PMID 30086778